CLINICAL TRIAL: NCT02607488
Title: Perioperative Systemic Lidocaine for Enhanced Bowel Recovery After Laparoscopic Bariatric Surgery: A Dose Dependent Study
Brief Title: Perioperative Systemic Lidocaine for Enhanced Bowel Recovery After Bariatric Surgery
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No fund no enough recruiting centers
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R-15-10-47
Record Dates: First submitted 2015-11-15; First posted 2015-11-18 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: Obese patients; Undergoing bariatric surgery
MeSH Terms: conditions — Obesity | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Patients will receive an intravenous bolus of 0.1 mL/kg of saline 0.9% solution followed by a continuous infusion 0.1 mL/kg/h of Saline 0.9% which will be continued for 24 hours after surgery.
  Interventions: Drug: Placebo
- Lidocaine 1% (Active Comparator): Patients will receive an intravenous bolus of 0.1 mL/kg of lidocaine 1.5% solution followed by a continuous infusion 0.1 mL/kg/h of lidocaine 1% solution which will be continued for 24 hours after surgery.
  All medications in the study protocol will be based on the dosing body weight [ideal body weight (IBW) + 0.4 × (actual body weight-IBW)]
  Interventions: Drug: Lidocaine 1%
- Lidocaine 1.5% (Active Comparator): Patients will receive an intravenous bolus of 0.1 mL/kg of lidocaine 1.5% solution followed by a continuous infusion 0.1 mL/kg/h of lidocaine 1,5% solution which will be continued for 24 hours after surgery.
  Interventions: Drug: Lidocaine 1.5%
- Lidocaine 2% (Active Comparator): Patients will receive an intravenous bolus of 0.1 mL/kg of lidocaine 1.5% solution followed by a continuous infusion 0.1 mL/kg/h of lidocaine 2% solution which will be continued for 24 hours after surgery.
  Interventions: Drug: Lidocaine 2%

INTERVENTIONS:
Drug: Placebo — Participants will receive an intravenous bolus of 0.1 mL/kg of saline 0.9% solution followed by a continuous infusion 0.1 mL/kg/h of Saline 0.9% which will be continued for 24 hours after surgery.
  All medications in the study protocol will be based on the dosing body weight [ideal body weight (IBW) + 0.4 × (actual body weight-IBW)]
  Arms: Placebo
Drug: Lidocaine 1% — Participants will receive an intravenous bolus of 0.1 mL/kg of lidocaine 1.5% solution followed by a continuous infusion 0.1 mL/kg/h of lidocaine 1% solution which will be continued for 24 hours after surgery.
  All medications in the study protocol will be based on the dosing body weight [ideal body weight (IBW) + 0.4 × (actual body weight-IBW)]
  Arms: Lidocaine 1%
Drug: Lidocaine 1.5% — Participants will receive an intravenous bolus of 0.1 mL/kg of lidocaine 1.5% solution followed by a continuous infusion 0.1 mL/kg/h of lidocaine 1.5% solution which will be continued for 24 hours after surgery.
  All medications in the study protocol will be based on the dosing body weight [ideal body weight (IBW) + 0.4 × (actual body weight-IBW)]
  Arms: Lidocaine 1.5%
Drug: Lidocaine 2% — Participants will receive an intravenous bolus of 0.1 mL/kg of lidocaine 1.5% solution followed by a continuous infusion 0.1 mL/kg/h of lidocaine 2% solution which will be continued for 24 hours after surgery.
  All medications in the study protocol will be based on the dosing body weight [ideal body weight (IBW) + 0.4 × (actual body weight-IBW)]
  Arms: Lidocaine 2%

SUMMARY:
Increasing rates of obesity over the last few decades have led to growing demand for bariatric surgery, which may resulted in decreased comorbidities and improved patient outcomes. Laparoscopic bariatric surgery has several clinical benefits in terms of improved quality of analgesia, reduced pulmonary complications, enhanced recovery of bowel function, less immune suppression, and shortened duration of hospital stay than open laparotomies.

Some investigators reported delayed return of bowel function for approximately two days after laparoscopic bariatric surgery, despite it occurred one day earlier than after open laparotomy. This potentially can lengthen the duration of hospital stay after bariatric procedures. With the impeding cost of health care in the developing countries, safely reducing length of stay is essential.

Other investigators reported early return of bowel movements during the first postoperative day in 65% of patients undergoing laparoscopic gastric bypass surgery due to reduced morphine use with implementation of a multimodal analgesia strategy including ketorolac, and propoxyphene hydrochloride/acetaminophen.

Lidocaine was investigated in several studies for its use in multi-modal management strategies to reduce postoperative pain and opioid use and enhance recovery. A recent Cochrane review including 45 trials demonstrated that systemic administration of lidocaine was associated with reduced pain scores at most of 'early time points' in patients undergoing laparoscopic abdominal surgery (MD -1.14, 95% CI -1.51 to -0.78; low-quality evidence), shorter times to first flatus (MD -5.49 hours, 95% CI -7.97 to -3.00; low-quality evidence) and first bowel movement (MD -6.12 hours, 95% CI -7.36 to -4.89; low-quality evidence), and less risk of paralytic ileus (risk ratio (RR) 0.38, 95% CI 0.15 to 0.99; low-quality evidence). However, no evidence of effect was found for lidocaine on shortening the time to first defecation. This low-quality evidence may be related to the heterogeneity between the studies in respect to the optimal dose, timing and duration of the administration of intravenous lidocaine.

DETAILED DESCRIPTION:
Hypothesis

Recognizing the need for enhanced bowel recovery for patients undergoing laparoscopic bariatric surgery, the investigators hypothesize that perioperative administration of low rather than high intravenous infusion rates of lidocaine can achieve early postoperative restoration of bowel motility at lower plasma levels.

Up to the best of the investigators' knowledge there is no study addressed the effects of perioperative administration of systemic lidocaine on postoperative recovery of bowel function in morbidly obese patients undergoing laparoscopic bariatric procedures.

Aim of the study

This trial aims to compare the effects of perioperative administration of escalating doses of intravenous lidocaine (1.0, 1.5 and 2.0 mg/kg/h) on the perioperative changes in hemodynamic, pain scores, and plasma lidocaine concentrations, postoperative recovery of bowel function, cumulative morphine use, hospital length of stay, and lidocaine related adverse effects in obese patients undergoing laparoscopic bariatric surgeries under general anesthesia.

Randomization

Five minutes before induction of general anesthesia, participants will be allocated randomly into four groups by drawing sequentially numbered sealed opaque envelopes containing a software-generated randomization code to receive an intravenous bolus of 0.1 mL/kg of either saline 0.9% or lidocaine 1.5% solution followed by a continuous infusion 0.1 mL/kg/h of Saline 0.9% or lidocaine 1%, 1.5% or 2% solution which will be continued for 24 hours after surgery. All medications in the study protocol will be based on the dosing body weight [ideal body weight (IBW) + 0.4 × (actual body weight-IBW)]. All study solutions looked identical and will be prepared by a local pharmacy. All staff in the operating room will be unaware of patient allocation group.

Perioperative management

An independent anesthesiologist who will not be involved in the study will instruct the participants preoperatively about the use of patient controlled analgesia and visual analogue scale to assess the severity of postoperative pain (0 mm for no pain and100 mm for worst imaginable pain).

Anesthetic management will be standardized. Oral ranitidine 150 mg and metoclopramide 10 mg will be administered the night before and 60 min before arrival in the operating room and subcutaneous enoxaparin 60 mg will be administered 12 h before the scheduled operation for prophylaxis against deep venous thrombosis.

Participant's monitoring includes electrocardiography, non-invasive blood pressure, pulse oximetry, plethysmography variability index (PVI) and capnography.

Following pre-oxygenation, in all participants, anesthesia will be induced with fentanyl 2-3 ug/kg and propofol 1.5-2.5 mg/kg. Rocuronium 0.6 mg/kg will be administered to facilitate tracheal intubation. Anesthesia will be initially maintained with 0.7-1.2 minimum alveolar concentrations (MAC) of sevoflurane in combination with air (1 L/min) and oxygen (1 L/min) mixture to maintain the mean arterial blood pressure (MAP) and heart rate (HR) are ≤20% of the baseline values. Fentanyl 0.5 ug/kg increments will be administered when the MAP and HR are ≥20% of the baseline values despite a MAC of sevoflurane ≥1.0. Rocuronium 0.1 mg/kg, will be used to maintain surgical relaxation.

Lungs will be initially ventilated in pressure-controlled mode to deliver a tidal volume of 8 ml/kg of predicted body weight (0.919 × (height in cm - 152.4) + 45.5 for women or 50 for men) at an I/E ratio of 1:2 and a positive end-expiratory pressure (PEEP) of 5 cmH2O. Respiratory rate will be adjusted to maintain end-tidal carbon dioxide tension (ETCO2) between 35 and 40 mm Hg.

All operations will be performed by the same surgeons. During CO2 pneumoperitoneum, the intra-abdominal pressure will be maintained at 12-14 mm Hg.

Participants position will be changed from supine to a 40° reverse Trendelenburg position.

During the operation, intraoperative fluid management was guided by a goal directed therapy algorithm using the PVI to guide fluid responsiveness. Hemodynamic control is standardized according to the investigators' protocol. Hypotension (defined as MAP value <25% of the baseline value on two consecutive readings within 3 min), not responding to decrease the sevoflurane MAC to 0.7 and a 5 ml/kg mL Ringer lactate or Acetate bolus over 5 min, will be treated with intravenous boluses of ephedrine, 3 mg or norepinephrine, 5 ug IV. Hypertension (defined as >20% increase in mean baseline MAP) will be treated by deepening anesthesia and administering doses of fentanyl, or labetalol, 20 mg. Tachycardia (defined as >20% increase in mean baseline HR) will be treated with esmolol, 20 mg. Bradycardia (HR <45) persisting for >2 min will be treated with glycopyrrolate, 0.2 mg IV, boluses.

Intravenous ondansetron, 4 mg IV, will be given for all participants for prevention of postoperative nausea and vomiting. Before wound closure, bupivacaine 0.25% will be infiltrated at all portals, and residual neuromuscular block will be antagonized with neostigmine, 50 µg/kg IV, and glycopyrrolate, 10 µg/kg IV. After completing surgery, sevoflurane will be discontinued and infusion of study medication will be continued for 24 h after the wound closure. Times from discontinuation of sevoflurane to eye opening, obeying simple commands (e.g., open mouth, squeeze hand) and tracheal extubation will be recorded.

Postoperative analgesic regime will be standardized in all participants including 30 mg of intravenous ketorolac every 6 h and paracetamol 1 g IV every 6 h and rescue doses of intravenous meperidine 25 mg. Participants will be discharged from the post-anesthesia care unit when they have a modified Aldrete score levels.

Intravenous fluids will run at 40 mL/h on the night of surgery and will be discontinued 24 h after surgery. Little attention is paid to urine output or oliguria in the absence of abnormal vital signs. Strict parameters for fluid boluses the night of surgery are in place based on hypotension and tachycardia. Active bedside mobilisation will be enforced for the first time the evening after surgery and assisted ambulation the morning after surgery at least twice a day.

Criteria for hospital discharge are as follows: absence of nausea and vomiting in the last 24 h, return of bowel function (daily defecation) and toleration of full diet, no to minimal pain (VAS less than 4), afebrile and no surgically associated morbidity (fever, wound dehiscence, wound infection, anastomotic leak, abscess). These variables will be recorded by a blind assessor to the allocation, every day at 10:00, 14:00 and 18:00 h. Patients ready for discharge after 14:00 h will be discharged on the following morning. All drains have to be removed before discharge.

Blindness

All staff in the operating room will be unaware of patient allocation group. Patients will be unaware about their allocation group. All study solutions looked identical and will be prepared by a local pharmacy.

Caregivers: An independent anesthesiologist who will not be involved in the study will instruct the patients preoperatively about the use of patient controlled analgesia and visual analogue scale to assess the severity of postoperative pain (0 mm for no pain and100 mm for worst imaginable pain) and will give the anesthetics and will be instructed to avoid using local anesthetics. An independent investigator involved in the assessment of the data and participants will be blind to the group assignment.

Statistical analysis:

Data will be tested for normality using the KolmogorovSmirnov test. Repeated-measures analysis of variance will be used for serial changes in the continuous data at different times after administration of study solution and the differences will be then corrected by post-hoc Bonferroni correction test. Fisher's exact test will be used for categorical data. Kruskal-Wallis one-way ANOVA and post-hoc Wilcoxon rank sum t-tests will be used for comparisons of the non-continuous data. Categorical data will be expressed as number (%), ordinal data will be expressed as median [range] and continuous data will be expressed as mean ± SD. A value of P<0.05 is considered to represent statistical significance.

Power analysis and sample size calculation:

Based on a previous study, the time to the return of bowel movements after laparoscopic bariatric surgery was normally distributed with a mean of 70 hours and a standard deviation of 22 hours. An a priori analysis indicated that 45 patients in each group would be sufficient to detect a 20% reduction in mean time to return of bowel movements, with a type I error of 0.005 (0.05/10 possible comparisons) and a power of 80%. The investigators added 15% more patients to account for drop-outs during the study.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients with a body mass index equal or greater than 35 kg/m2.
* American Society of Anesthesiologists (ASA) II-III
* Patients scheduled for laparoscopic bariatric surgery under general anesthesia

Exclusion Criteria:

* History of significant cardiac disease.
* History of significant respiratory disease.
* History of significant hepatic disease.
* History of significant renal diseases.
* History of an atrio-ventricular block grade II to III.
* Long QT syndrome.
* Pre-existing disorder of the gastrointestinal tract.
* Patients with history of alcohol or drug abuse.
* Allergy to amide local anesthetics.
* History of epilepsy.
* Pregnancy.
* Patients receiving cardiovascular medications.
* Patients receiving steroids.
* Patients receiving an opioid analgesic medication within 24 h before the operation.
* Conversion from a laparoscopic to an open laparotomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative recovery of bowel function | For 72 hours after surgery
  Times to first passage of flatus, first defecation, and tolerating liquids measured in hours from the end of surgery. Patients will be asked to note the time they will be able to tolerate liquids and their first passage of flatus ("gas").

SECONDARY OUTCOMES:
Perioperative changes in heart rate | For 48 hours after surgery
  Heart rate will be recorded before induction of anesthesia, 5 min after induction, every 15 min intraoperatively, and then 1 h, 4 h, 12 h, 24 h, 36 h, 48 h after surgery
Perioperative changes in blood pressure | For 48 hours after surgery
  Blood pressure will be recorded before induction of anesthesia, 5 min after induction, every 15 min intraoperatively, and then 1 h, 4 h, 12 h, 24 h, 36 h, 48 h after surgery
Pain scores | For 48 hours after surgery
  Four-hourly pain scores at rest and during movement and cough
Intraoperative total use of fentanyl | For 4 hours after induction of anaesthesia
  Fentanyl0.5 micrograms/kilogram of body weight will be administered intravenously on the discretion of the charged anesthesiologist in case of inadequate intraoperative analgesia
Perioperative use of intravenous fluids | For 48 hours after surgery
  The volume of intravenously administered fluid therapy will be recorded before, during, and after surgery.
Perioperative use of norepinephrine | For 48 hours after surgery
  The volume of intravenously administered norepinephrine to treat low blood pressure will be recorded before, during, and after surgery.
Perioperative use of dobutamine | For 48 hours after surgery
  The volume of intravenously administered dobutamine to treat low cardiac output will be recorded before, during, and after surgery.
The balance between the fluid intake and output | For 48 hours after surgery
  The balance between the fluid intake and output during surgery and 34 hours and 48 hours after surgery will be recorded
Postoperative cumulative morphine use | For 48 hours after surgery
  Intravenous morphine will be administered intravenously as per request of the participants to relief their postoperative pain. The cumulative consumption of morphine by participants will be recorded at 24 hours and 48 hours after surgery
Times to clinical recovery | For 2 hours after surgery
  Times to spontaneous breathing, eye opening, obeying verbal commands, and extubation
Length of Post-Anaesthesia Care Unit stay | For 4 hours after surgery
Time to readiness for hospital | for 10 days after surgery
Time to actual discharge from hospital | For 10 days after surgery
Perioperative changes in cognitive function | For 48 hours after surgery
  It will be assessed using as assessed by a mini mental score preoperatively (baseline) and 24 h and 48 h after surgery
Overall patient satisfaction score | For 48 hours after surgery
  This will be assessed using a 100-point scale with 1 = completely dissatisfied to 100 = completely satisfied) will be recorded on postoperative day (POD)s 1, and 2
Postoperative nausea and vomiting | For 48 hours after surgery
  It will be scored 4-hourly as follows; (0: no nausea; 1: nausea no vomiting; 2: nausea and vomiting)
Postoperative pruritus | For 48 hours after surgery
  This will be assessed at four hourly as follows pruritus rated using a categorical scale (0, none; 1, mild; 2, moderate; and 3, severe)
Postoperative sedation | For 48 hours after surgery
  This will be assessed at 4-hourly using sedation score (four-point verbal rating scores (VRS): awake, drowsy, arousable or deep sleep)
Number of participants with surgery-related complications | For 15 days after surgery
  These include the occurrence of bleeding, fever, wound dehiscence, wound infection, anastomotic leak, abscess, peritonitis, infection
Associated comorbidities | For 1 day before induction of anaesthesia
  These include preoperative diabetes, renal impairment, hepatic dysfunction, cardiac dysfunction, pulmonary disease, endocrine disease
Number of participants with lidocaine treatment-related adverse events | For 48 hours after surgery
  These adverse events include arrhythmia, sedation, nausea and vomiting, light-headedness, headache, perioral numbness, tunnel vision, or seizures
Serum lidocaine level | For 48 hours after surgery
Plasma albumin level | For 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, MD, Study Chair — Departments of Anaesthesia and Surgical Intensive Care, College of Medicine, Mansoura University, Egypt, and Anesthesiology Department, College of Medicine, University of Dammam, Saudi Arabia; Samah El Kenany, MD, Principal Investigator — Department of Anaesthesia and Surgical Intensive Care, College of Medicine, Mansoura University, Egypt
Locations (1):
- Mansoura University Hospitals, Al Mansurah, DK, Egypt